CLINICAL TRIAL: NCT00420498
Title: Effects of Atomoxetine on Cognitive Function in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27678; NARSAD
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia; Cognition; Smoking
Keywords: Schizophrenia; Prefrontal Cortical Function; Smoking; Cognition; Positive and Negative Symptoms; Tobacco; Cigarette Smoking; Dopamine
MeSH Terms: conditions — Schizophrenia; Smoking; Cigarette Smoking | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atomoxetine (Strattera™)

SUMMARY:
The purpose of this study is to examine the effects of atomoxetine (Strattera™) on prefrontal cognitive functioning in persons with schizophrenia. Secondarily, the effects of atomoxetine on positive and negative symptoms and on cigarette smoking consumption in persons with schizophrenia will be examined.

DETAILED DESCRIPTION:
Schizophrenia occurs in approximately 1% of the general population. Hallmark symptoms of schizophrenia include positive and negative symptoms, as well as deficits in various aspects of cognitive function, with particular reference to neuropsychological tasks related to the prefrontal cortex (PFC). A leading theory with respect to these deficits in prefrontal cortical functioning is that there is dysregulation (with overall hypofunction) of mesocortical dopamine (DA) projections from the VTA to the prefrontal cortex (PFC) in persons with schizophrenia, thus diminishing abilities on tasks mediated by these cortical areas [1]. Further, it is thought that the high rates of smoking in schizophrenia (58-88%) as compared to a non-psychiatric population (~25%) may be due in part to the tendency of schizophrenic patients to remediate these neurocognitive deficits by cigarette smoking, as nicotine has been shown to improve selected cognitive deficits in persons with this illness [2-4], and in fact such cognitive deficits may be a vulnerability factor predisposing these patients to initiate and maintain smoking [5].

Atomoxetine (Strattera™) which has efficacy in treating children and adults with Attention Deficit Hyperactivity Disorder (ADHD). It increases extracellular levels of both NE and DA in the PFC by blocking the NE transporter (NET), where it has been shown that DA is predominately taken up non-selectively by NET [6]. In contrast, atomoxetine was not found to increase extracellular DA in subcortical areas [6]. It can be theorized that atomoxetine may selectively increase DA in the PFC (versus subcortical areas) by inhibition of NETs in the PFC. Accordingly, since persons with schizophrenia are thought to have a deficit of DA in the PFC, and excessive subcortical DA function, a NET inhibitor such as atomoxetine may increase DA-dependent PFC-mediated neurocognitive functioning, and reduce negative symptoms associated with this disorder, without worsening positive symptoms of schizophrenia. Atomoxetine has been shown to be safe and effective for ADHD treatment in both children and adults (Eiland, 2004). Little is known about Atomoxetine's effects in treating other psychiatric disorders, however, it has been hypothesized that this medication may have efficacy for cognitive remediation in the schizophrenic population (Friedman, 2004).

In order to more fully understand the effects of this medication, a double-blind, placebo-controlled clinical trial is proposed in which sixty (60) participants with schizophrenia who are cigarette smokers would be randomized in a double-blind manner to one of three doses of atomoxetine [0.0 mg/day (n=20) , 40.0 mg/day (n=20), or 80.0 mg/day (n=20)]. Doses were chosen in accordance with the FDA suggested dosing, including a schedule of initiation starting with 40.0mg/day and a target recommended dose of 80.0mg/day which may be reached within a three day period. The highest recommended dose is 100 mg/day. These doses were ultimately selected for this study because they are doses that are believed to be well-tolerated by patients, doses that may be achieved within the two-week period of this study, and two doses that fit with our intention to study the dose-dependent effects of this medication. Safety and effectiveness for these doses has been determined for patients 18 years of age and older with ADD, the population that has been studied using Atomoxetine. Should we discover that our patients with schizophrenia do not tolerate these doses well through extensive monitoring of their physiological and clinical symptoms, or that the maximum dose of 80.0 mg/day cannot be reached during this time period, smaller doses will be considered and the appropriate amendments will be submitted.

Participants would be assessed across three cognitive testing sessions over a two-week period including baseline assessments Day 1 (prior to medication administration), on Day 8 (after one week of medication), and again on Day 15 (after two weeks of medication). No data currently exists in the literature regarding specific improvements in neurocognitive performance in schizophrenia with atomoxetine, although it has been hypothesized that this medication may be specifically helpful in schizophrenia. Therefore we believe this will be one of the first studies of its kind. We hypothesize that atomoxetine will dose-dependently improve deficits in PFC-related cognitive performance in persons with schizophrenia. We secondarily hypothesize that schizophrenic smokers will demonstrate a reduction in negative symptoms and daily cigarette consumption with atomoxetine as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 and 59;
* SCID-I for DSM-IV diagnosis of schizophrenia or schizoaffective disorder, and nicotine dependence
* Smoking at least 15 cigarettes per day, and have expired breath CO level >10 ppm,
* Be in stable remission from active psychiatric symptomatology, (as judged by trained clinical staff in the PRISM research program) and be on a stable dose of psychiatric medication(s) for the past 3 months
* No current abuse or dependence of alcohol or other substances of abuse within the past 3 months,
* Full scale IQ > 80,
* Presence of definable cognitive deficits of interest including VSWM, CPT, and WCST (e.g. at least one standard deviation below average).
* Able to give informed consent for participation.

Exclusion Criteria:

* Meet DSM-IV criteria for other major Axis I disorders besides those specified for each diagnostic group.
* Current abuse or dependence of alcohol or substances within the last 3 months, and subjects who are methadone maintained will be excluded.
* Full scale IQ < 80.
* Unable to give informed consent.
* Patients who are pregnant or planning on becoming pregnant will not be included in this study.
* Patients on paroxetine, fluoxetine, and quinidine will be excluded from this study.
* Are deemed medically unsafe to take atomoxetine, as judged by the study physician. Contraindications to the use of atomoxetine include hypersensitivity to atomoxetine, concurrent use of monoamine oxidase inhibitors (atomoxetine should be avoided during therapy with or within 2 weeks of discontinuing an MAO inhibitor), and patients with narrow angle glaucoma. Precautions would include concomitant administration with CYP 2D6 inhibitors (eg, paroxetine, fluoxetine, quinidine) (which would necessitate a dose adjustment with atomoxetine), liver disease (enhanced risk of toxicity; empiric dose reduction is suggested based on clinical response; the drug should be avoided in acute hepatic failure), patients with hypertension, tachycardia, or other cardiovascular or cerebrovascular disease, patients with or at risk of hypotension , patients with urinary retention or bladder dysfunction.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To examine the effects of atomoxetine (Strattera™) on prefrontal cognitive functioning in persons with schizophrenia.

SECONDARY OUTCOMES:
To examine the effects of atomoxetine on positive and negative symptoms and on cigarette smoking consumption in persons with schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi A Sacco, Psy.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, SAC-115, New Haven, Connecticut, United States